CLINICAL TRIAL: NCT02085850
Title: Incidence and Progression of Glaucoma in the Tema Eye Survey Cohort
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tema Christian Eye Center (Other)
Responsible Party: Principal Investigator, Alex Spratt, Principal Investigator, Tema Christian Eye Center
Other Study IDs: TCEC 066/13-14
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects identified in the Tema Eye Survey: Subjects identified in the Tema Eye Survey

SUMMARY:
Aim 1: To determine the incidence of glaucoma in Ghana in subjects previously found to be non-glaucomatous in the Tema Eye Survey.

Aim 2: To characterise the progression of glaucoma and the outcomes of subjects diagnosed with glaucoma in the Tema Eye Survey.

ELIGIBILITY:
Inclusion Criteria:

- glaucomatous and non-glaucomatous patients previously seen in the Tema Eye Survey who are selected and invited to participate

Exclusion Criteria:

- patients not previously seen in the Tema Eye Survey

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 1375 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Glaucoma | Day 0
Progression of Glaucoma | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Spratt, MBBCh FRCOphth, Principal Investigator — Tema Christian Eye Center; Donald L Budenz, MD MPH, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- Tema Christian Eye Center, Tema, Ghana